CLINICAL TRIAL: NCT00846755
Title: Impact of Treating Thyroid Hormone Dysfunction During Pregnancy: A Randomized Controlled Trial of Universal Screening Versus Case Finding
Brief Title: Thyroid Disease in Pregnancy: Case Finding Versus Universal Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale V. Fazzi (Other)
Responsible Party: Principal Investigator, Dr. Roberto Negro, MD, Ospedale V. Fazzi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LE-1126-IT
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-09

CONDITIONS: Thyroid Disease; Pregnancy
Keywords: Thyroid; Pregnancy
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyroxine; Propylthiouracil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Levothyroxine, Propylthiouracil (Active Comparator): Drugs for the treatment of thyroid disease, are administered, when necessary, in high risk women, either in case finding, or in Universal Screening Group
  Interventions: Drug: Levothyroxine, Propylthiouracile
- clinical checks (No Intervention): Low risk women whose sera are tested postpartum. Then patients with undiagnosed thyroid disease, are not treated

INTERVENTIONS:
Drug: Levothyroxine, Propylthiouracile — Drugs were titrated to render euthyroid pregnant patients with thyroid disease
  Other Names: Levothyroxine; Propylthiouracile
  Arms: Levothyroxine, Propylthiouracil

SUMMARY:
The purpose of this study is to determine whether treatment of thyroid disease during pregnancy decrease the incidence of adverse outcome, and to compare the impact of Universal Screening versus case Finding strategy in detecting thyroid dysfunction

DETAILED DESCRIPTION:
Thyroid disease during pregnancy has been associated with multiple adverse outcomes including miscarriage, preterm delivery, postpartum thyroiditis and decreased IQ in the offspring. Whether or not all women should be screened for thyroid disease during pregnancy (Universal Screening), screening should be confined to women at high risk for thyroid disease (Case Finding), or no screening should occur is controversial. For this purpose, pregnant women in the first trimester are randomly assigned to the Screening group or Case finding group. All women in the Screening group and high-risk women in the Case Finding group are immediately tested for FT4, TSH and TPO antibodies. Low-risk women in the Case Finding group have their sera tested postpartum. levothyroxine or PTU are given in hypothyroid and hyperthyroid women respectively. Outcome Measure: total number of adverse events occurring during pregnancy and in the neonatal period controlling for clustering of outcomes within women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Within 11 week of gestation

Exclusion Criteria:

* Already known thyroid disease

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4657 (Actual)
Dates: Start 2005-03; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
number of adverse outcomes which occur during pregnancy and in the neonatal period in patients divided in Case Finding and Universal Screening groups | 9 months

SECONDARY OUTCOMES:
Evaluation of the efficacy of Case Finding and Screening strategy | 4 years
Intelligence Quotient | 6 years
  •Intellectual function of children at 6 years of age, as measured by the Wechsler Intelligence Scale for Children (WISC) III, in women with a)hypothyroidism, left untreated because belonging to Case Finding Low Risk Group, b) hypothyroidism, treated with levothyroxine because belonging to Universal Screening High Risk and Low Risk Groups, and in Case Finding High Risk Group, and c)euthyroidism (control group)

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Negro, Dr, Principal Investigator — "V. Fazzi" Hospital
Locations (1):
- "V. Fazzi" Hospital, Lecce, Italy

REFERENCES:
- [Derived] Negro R, Schwartz A, Gismondi R, Tinelli A, Mangieri T, Stagnaro-Green A. Thyroid antibody positivity in the first trimester of pregnancy is associated with negative pregnancy outcomes. J Clin Endocrinol Metab. 2011 Jun;96(6):E920-4. doi: 10.1210/jc.2011-0026. Epub 2011 Mar 16. PMID 21411559
- [Derived] Stagnaro-Green A, Schwartz A, Gismondi R, Tinelli A, Mangieri T, Negro R. High rate of persistent hypothyroidism in a large-scale prospective study of postpartum thyroiditis in southern Italy. J Clin Endocrinol Metab. 2011 Mar;96(3):652-7. doi: 10.1210/jc.2010-1980. Epub 2010 Dec 29. PMID 21190974